CLINICAL TRIAL: NCT06394492
Title: A Randomized, Open-Label, Controlled, Phase III Study of SHR-A1921 Versus Investigator's Choice of Chemotherapy in Patients With Platinum-Resistant Recurrent Epithelial Ovarian Cancer
Brief Title: SHR-A1921 for Injection in Patients With Platinum-Resistant Recurrent Epithelial Ovarian Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1921-303
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Doxorubicin; Paclitaxel; Topotecan

STUDY DESIGN:
Intervention Model Description: To evaluate the efficacy and safety of SHR-A1921 compared with investigator-chosen chemotherapy in patients with platinum-resistant recurrent epithelial ovarian cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group 1: SHR-A1921 (Experimental)
  Interventions: Drug: SHR-A1921
- Treatment group 2: Investigator's choice of chemotherapy (Active Comparator)
  Interventions: Drug: Doxorubicin; Drug: Paclitaxel; Drug: Topotecan

INTERVENTIONS:
Drug: SHR-A1921 — SHR-A1921 dose 1
  Arms: Treatment group 1: SHR-A1921
Drug: Doxorubicin — Doxorubicin dose 2
  Arms: Treatment group 2: Investigator's choice of chemotherapy
Drug: Paclitaxel — Paclitaxel dose 3
  Arms: Treatment group 2: Investigator's choice of chemotherapy
Drug: Topotecan — Topotecan dose 4
  Arms: Treatment group 2: Investigator's choice of chemotherapy

SUMMARY:
This study is a randomized, open-label, controlled, phase III study to evaluate the efficacy and safety of SHR-A1921 versus investigator's choice of chemotherapy in patients with platinum-resistant recurrent epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent.
2. 18 years and older, female.
3. Pathologically diagnosed epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.
4. Patients must have platinum-resistant disease
5. Be able to provide fresh or archived tumour tissue.
6. At least one measurable lesion according to RECIST v1.1.
7. Eastern Cooperative Oncology Group (ECOG) score: 0-1.
8. With a life expectancy ≥ 12 weeks.
9. Adequate bone marrow reserve and organ function.
10. Contraception is required during the trial.

Exclusion Criteria:

1. Uncontrolled pleural effusion, pericardial effusion, or abdominal effusion with clinical symptoms.
2. Previous or co-existing malignancies.
3. Current or History of ILD.
4. Clinical symptoms or diseases of the heart that are not well controlled.
5. Arterial/venous thrombosis events occurred before the first dose.
6. Grade ≥2 bleeding events of CTCAE occurred before the first dose.
7. Gastrointestinal perforation or fistula, urethral fistula, abdominal abscess occurred before the first dose.
8. Patients with intestinal obstruction or parenteral nutrition before the first dose.
9. Serious infection before the first dose.
10. Active hepatitis B or active hepatitis C.
11. Received systemic anticancer treatments 4 weeks prior to the initiation of the study treatment.
12. Treated with TOP1 inhibitors or ADCs with TOP1 inhibitors as payload.
13. Unresolved CTCAE ≥grade 2 toxicities from previous anticancer therapy.
14. History of severe hypersensitivity reactions to either the drug substances or inactive ingredients of SHR-A1921.
15. Other inappropriate situation considered by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) assessed by Blinded Independ Review Committee (BIRC) as per RECIST 1.1 | Screening up to study completion, an average of 1 year

SECONDARY OUTCOMES:
Overall Survival (OS) | Screening up to study completion, an average of 1 year
Objective Response Rate (ORR), assessed by site investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Duration of Response (DoR), assessed by site investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Disease Control Rate (DCR), assessed by site investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year
Response Rate (RR) assessed by RECIST 1.1 and Gynaecologic Cancer Intergroup (GCIG) criteria | Screening up to study completion, an average of 1 year
CA-125 Response Rate assessed by the Gynaecologic Cancer Intergroup (GCIG) criteria | Screening up to study completion, an average of 1 year
Adverse Events | Screening up to study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - National Cancer Center/Tumor Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided